CLINICAL TRIAL: NCT00777140
Title: Double-blind, Randomized, Placebo Controlled, Dose-finding Phase 2 Clinical Trial of Intravenous Deferoxamine in Patients With Acute Ischemic Stroke Treated With Tissue Plasminogen Activator
Brief Title: Thrombolysis and Deferoxamine in Middle Cerebral Artery Occlusion
Acronym: TANDEM-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Principal Investigator, Monica Millan Torne, Medical Doctor, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TANDEM-1; EUDRACT: 2007-006731-31
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Ischemic Stroke, Acute
Keywords: Stroke; Ischemic Stroke; Thrombolytic treatment; Middle cerebral artery occlusion; Deferoxamine; Iron chelator; Acute Ischemic Stroke treated with Intravenous Thrombolytic
MeSH Terms: conditions — Ischemic Stroke; Stroke; Infarction, Middle Cerebral Artery | interventions — Deferoxamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1. Deferoxamine (Active Comparator): Intravenous deferoxamine: bolus of 10mg/Kg (initiated during tPA infusion) and perfusion of 20/40/60 mg/Kg/day during 72h. Three different doses (3 steps), 15 patient in the active arm for each dose.
  Interventions: Drug: Deferoxamine
- 2. Placebo (Placebo Comparator): Saline solution: Bolus and perfusion during 72h. 5 patients in the placebo arm in each step (randomization 3:1)
  Interventions: Drug: Deferoxamine

INTERVENTIONS:
Drug: Deferoxamine — Intravenous deferoxamine: bolus 10mg/Kg (initiated during thrombolytic infusion, iv tPA), followed by intravenous perfusion of 20/40/60mg/Kg during 72h. It's a dose-finding study with 3 different doses of deferoxamine, with 20 patients (15 active:5 placebo) in each step.
  Bolus + 72h perfusion of saline solution for the placebo group.

SUMMARY:
Iron overload has been associated with greater brain injury in ischemia/reperfusion experimental stroke models and ischemic stroke patients, especially in those treated with thrombolytic treatment. Deferoxamine administration, an iron chelator, offers a neuroprotective action in ischemia/reperfusion animal models.

Primary objective: To evaluate the security and tolerability of deferoxamine endovenous treatment in acute ischemic stroke patients treated with iv. tPA.

Secondary objectives: To study pharmacokinetics of deferoxamine given by endovenous bolus (10 mg/Kg) followed by 72-hour continuous intravenous infusion (20, 40 o 60 mg/Kg). To evaluate the deferoxamine effect in clinical outcome, infarct volume and hemorrhagic transformation and brain edema development.

Methodology: Double-blind, randomized, placebo controlled, dose-finding phase II clinical trial. Study stages: 1st: bolus+20 mg/Kg/day vs. Placebo (n=15:5); 2nd: bolus+40 mg/Kg/day vs. Placebo (n=15:5); 3rd: bolus+60 mg/Kg/day vs placebo (n=15:5). These doses will be increased according to security results of the previous stage. Patients will be continuously monitored in stroke units. Laboratory parameters will be measured at baseline, 24h, 72h and 30 days to evaluate adverse events related to the drug. Serum deferoxamine and feroxamine concentrations will be measured along time after the injection in a subgroup of patients to the pharmacokinetics study. CT scan will be performed at 24-36h to assess hemorrhagic transformation and brain edema. The NIH Stroke Scale will be evaluated during hospitalization, and the Rankin score at discharge and 3 months.

If deferoxamine demonstrate to be secure and well tolerated treatment in acute stroke patients, it may be a new therapy option to lower the brain injury after ischemia and reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old
* Acute Ischemic Stroke on the middle cerebral artery territory
* Treatment with iv tPA in the first 3 hours from symptoms onset

Exclusion Criteria:

* Modified Rankin Scale more or equal to 2
* Infectious, inflammatory, neoplastic or hematologic disease
* Anemia (Hto<34% or Hb<10g/dl)
* Previous renal failure
* Previous treatment with oral iron supplement
* Minor stroke (NIHSS less than 4), lacunar or posterior territory
* Alcohol consumption (more than 40mg/Kg)
* Pregnancy
* Participation in other clinical trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Clinical and Analytical Adverse Events (anemia, hypotension, renal failure, mortality, hemorrhagic transformation, cerebral edema, other severe adverse events) | 3 months

SECONDARY OUTCOMES:
Neurological status (NIHSS, Barthel and Rankin scales), final ischemic lesion volume on CTscan. | 24h, 7days and 3 months
Deferoxamine and ferritin levels in serum (pharmacokinetics). | 72h

CONTACTS AND LOCATIONS:
Overall Officials: Monica Millán Torné, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (4):
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, La Coruña, Galicia
  - Hospital Universitari Josep Trueta, Girona
  - Hospital Universitario de la Princesa, Madrid

REFERENCES:
- [Background] Kontos HA. Oxygen radicals in cerebral ischemia: the 2001 Willis lecture. Stroke. 2001 Nov;32(11):2712-6. doi: 10.1161/hs1101.098653. PMID 11692043
- [Background] Selim MH, Ratan RR. The role of iron neurotoxicity in ischemic stroke. Ageing Res Rev. 2004 Jul;3(3):345-53. doi: 10.1016/j.arr.2004.04.001. PMID 15231241
- [Background] Castellanos M, Puig N, Carbonell T, Castillo J, Martinez J, Rama R, Davalos A. Iron intake increases infarct volume after permanent middle cerebral artery occlusion in rats. Brain Res. 2002 Oct 11;952(1):1-6. doi: 10.1016/s0006-8993(02)03179-7. PMID 12363398
- [Background] Millan M, Sobrino T, Castellanos M, Nombela F, Arenillas JF, Riva E, Cristobo I, Garcia MM, Vivancos J, Serena J, Moro MA, Castillo J, Davalos A. Increased body iron stores are associated with poor outcome after thrombolytic treatment in acute stroke. Stroke. 2007 Jan;38(1):90-5. doi: 10.1161/01.STR.0000251798.25803.e0. Epub 2006 Nov 30. PMID 17138950
- [Background] Davalos A, Castillo J, Marrugat J, Fernandez-Real JM, Armengou A, Cacabelos P, Rama R. Body iron stores and early neurologic deterioration in acute cerebral infarction. Neurology. 2000 Apr 25;54(8):1568-74. doi: 10.1212/wnl.54.8.1568. PMID 10762495
- [Background] Davalos A, Fernandez-Real JM, Ricart W, Soler S, Molins A, Planas E, Genis D. Iron-related damage in acute ischemic stroke. Stroke. 1994 Aug;25(8):1543-6. doi: 10.1161/01.str.25.8.1543. PMID 8042204
- [Background] Erdemoglu AK, Ozbakir S. Serum ferritin levels and early prognosis of stroke. Eur J Neurol. 2002 Nov;9(6):633-7. doi: 10.1046/j.1468-1331.2002.00472.x. PMID 12453079
- [Background] Soloniuk DS, Perkins E, Wilson JR. Use of allopurinol and deferoxamine in cellular protection during ischemia. Surg Neurol. 1992 Aug;38(2):110-3. doi: 10.1016/0090-3019(92)90087-4. PMID 1509342
- [Background] Patt A, Horesh IR, Berger EM, Harken AH, Repine JE. Iron depletion or chelation reduces ischemia/reperfusion-induced edema in gerbil brains. J Pediatr Surg. 1990 Feb;25(2):224-7; discussion 227-8. doi: 10.1016/0022-3468(90)90407-z. PMID 2303992
- [Background] Palmer C, Roberts RL, Bero C. Deferoxamine posttreatment reduces ischemic brain injury in neonatal rats. Stroke. 1994 May;25(5):1039-45. doi: 10.1161/01.str.25.5.1039. PMID 8165675
- [Background] Hurn PD, Koehler RC, Blizzard KK, Traystman RJ. Deferoxamine reduces early metabolic failure associated with severe cerebral ischemic acidosis in dogs. Stroke. 1995 Apr;26(4):688-94; discussion 694-5. doi: 10.1161/01.str.26.4.688. PMID 7709418
- [Background] Freret T, Valable S, Chazalviel L, Saulnier R, Mackenzie ET, Petit E, Bernaudin M, Boulouard M, Schumann-Bard P. Delayed administration of deferoxamine reduces brain damage and promotes functional recovery after transient focal cerebral ischemia in the rat. Eur J Neurosci. 2006 Apr;23(7):1757-65. doi: 10.1111/j.1460-9568.2006.04699.x. PMID 16623832
- [Background] Kim HJ, Hida H, Jung CG, Miura Y, Nishino H. Treatment with deferoxamine increases neurons from neural stem/progenitor cells. Brain Res. 2006 May 30;1092(1):1-15. doi: 10.1016/j.brainres.2006.02.046. Epub 2006 May 12. PMID 16697980
- [Background] Summers MR, Jacobs A, Tudway D, Perera P, Ricketts C. Studies in desferrioxamine and ferrioxamine metabolism in normal and iron-loaded subjects. Br J Haematol. 1979 Aug;42(4):547-55. doi: 10.1111/j.1365-2141.1979.tb01167.x. PMID 476006
- [Background] Allain P, Mauras Y, Chaleil D, Simon P, Ang KS, Cam G, Le Mignon L, Simon M. Pharmacokinetics and renal elimination of desferrioxamine and ferrioxamine in healthy subjects and patients with haemochromatosis. Br J Clin Pharmacol. 1987 Aug;24(2):207-12. doi: 10.1111/j.1365-2125.1987.tb03163.x. PMID 3620295
- [Derived] Millan M, DeGregorio-Rocasolano N, Perez de la Ossa N, Reverte S, Costa J, Giner P, Silva Y, Sobrino T, Rodriguez-Yanez M, Nombela F, Campos F, Serena J, Vivancos J, Marti-Sistac O, Cortes J, Davalos A, Gasull T. Targeting Pro-Oxidant Iron with Deferoxamine as a Treatment for Ischemic Stroke: Safety and Optimal Dose Selection in a Randomized Clinical Trial. Antioxidants (Basel). 2021 Aug 10;10(8):1270. doi: 10.3390/antiox10081270. PMID 34439518
- [Derived] Van der Loo LE, Aquarius R, Teernstra O, Klijn K, Menovsky T, van Dijk JMC, Bartels R, Boogaarts HD. Iron chelators for acute stroke. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD009280. doi: 10.1002/14651858.CD009280.pub3. PMID 33236783